CLINICAL TRIAL: NCT04359524
Title: Fitness and Health Characteristics in Conscripts With Supplementation of Vitamin D
Brief Title: Vitamin D Supplementation in Conscripts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leho Rips (Other)
Collaborators: Estonian Defence Forces (Unknown); University of Tartu (Other)
Responsible Party: Sponsor-Investigator, Leho Rips, Head of department, Tartu University Hospital
Organization: Tartu University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R-002
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Vitamin D Deficiency; Military Activity
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Triple blinded randomized placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Computed randomization was used to divide conscripts into two groups; either the intervention group, who received vitamin D3 capsules (1200 IU/30µg) or the control group, who received placebo (oil capsules).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Received vitamin D3 capsules (1200 IU/30µg).
  Interventions: Dietary Supplement: Vitamin D3 (1200 IU/30µg)
- Control (Placebo Comparator): Received placebo (oil capsules).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (1200 IU/30µg)
  Arms: Intervention
Dietary Supplement: Placebo — Placebo oil capsule
  Arms: Control

SUMMARY:
A longitudinal, triple-blinded, randomized, placebo-controlled trial, with a 7-month follow-up period is conducted between October 2016 to April 2017.

DETAILED DESCRIPTION:
Body mass (kg) and height (cm) is measured by the same person at the medical center using standardized equipment and the body mass index (BMI) is calculated in kg/m2.

Computed randomization is used to divide conscripts into two groups; either the intervention group or the control group. Both types of capsules are administered once per day in the morning before breakfast for 7 months. Standardized coded packages (3 per conscript) and capsules (100 per package) are manufactured on a special order by Innopharma A/S (Denmark). No commercial sponsoring is involved.

The key of the package code is stored in the computer database until unblinding of the results.

Laboratory measurements Serum samples for clinical chemistry analysis are collected into serum clot activator tubes. Calcium measurements are performed using spectrophotometry method. Ionized calcium measurements are performed using ion selective electrodes. The direct chemiluminescent immunoassay method is used for measurement of PTH. 25(OH)D is measured using direct chemiluminescent immunoassay method.

Power calculation The primary variable of the study is the level of 25 (OH)D in the serum. In the power analysis a difference of 20 nmol/L between the intervention and the control group is considered to be meaningful to detect. If the SD would be 25 nmol/L, then 26 participants would be needed in each group to reach a power of 80%.

Statistical analysis The distribution of blood serum values in the study groups is described by means and standard deviations (SD). Differences in mean values of the variables of interest between the groups are evaluated using Welch t-test. The within group comparisons over time are performed using paired t-test with Bonferroni correction. Distributions of categorical variables are described by absolute numbers and percentages and compared between groups using the Fisher exact test. Statistical significance is set at the 0.05 probability level.

ELIGIBILITY:
Inclusion Criteria:

* participating in military service at the Estonian Defence Forces
* voluntarity to participate in the study

Exclusion Criteria:

* inability to continue military service for any reason, during the 7 month follow-up period

Ages: 19 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of vitamin D deficence | 0, 2, 5 and 7 months of recruitment
  Prevalence of vitamin D deficence as measured serum vitamin D 25(OH)D concentration. Vitamin D was considered as sufficient if the se-rum 25(OH)D concentration was ≥75 nmol/L, insufficient if <75 nmol/L, and deficient if <50 nmol/L.

OTHER OUTCOMES:
serum parathyroid hormone | 0, 2, 5 and 7 months of recruitment
  serum parathyroid hormone concentration (pmol/l)
serum calcium | 0, 2, 5 and 7 months of recruitment
  serum calcium (Ca) concentration (mmol/l)
serum ionized calcium | 0, 2, 5 and 7 months of recruitment
  serum ionized calcium (Ca-i) concentration (mmol/l)
Hand Grip Strength | 0, 2, 5 and 7 months of recruitment
  Hand grip strength is determined by isometric contraction while standing, upper limb away from the body, using a hand dynamometer (Lafayette Instrument Co., USA).
Testosterone | 0, 2, 5 and 7 months of recruitment
  Serum testosterone concentration (nmol/l)
Cortisol | 0, 2, 5 and 7 months of recruitment
  Serum cortisol concentration (nmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gapeyeva, MD, PhD, Study Director — University of Tartu
Locations (1):
- Kuperjanov Infantry Battalion, Estonian Defence Forces, Võru, Võrumaa, Estonia